CLINICAL TRIAL: NCT04514042
Title: Comparison of Zenker's Diverticulum Treatment Using Peroral Endoscopic Myotomy and Flexible Endoscopy Septotomy: International, Multicentre, Randomized, Double-blind Clinical Trial.
Brief Title: Comparison of Zenker's Diverticulum Treatment Using Peroral Endoscopic Myotomy and Flexible Endoscopy Septotomy.
Acronym: ZIPPY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Centre of Postgraduate Medical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3299445
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-03

CONDITIONS: Zenker Diverticulum; Diverticulum, Esophago-Pharyngeal; Diverticulum, Esophageal; Dysphagia; Gastrointestinal Disease
Keywords: Cricopharyngeus myotomy; Peroral endoscopic myotomy; Submucosal tunneling endoscopic septum division; Flexible endoscopy septotomy
MeSH Terms: conditions — Zenker Diverticulum; Diverticulum, Esophageal; Deglutition Disorders; Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard procedure (Active Comparator): Patients with Zenker's diverticulum treated with flexible endoscopy septotomy.
  Interventions: Procedure: Flexible endoscopic septotomy
- Investigational procedure (Experimental): Patients with Zenker's diverticulum treated with peroral endoscopic myotomy.
  Interventions: Procedure: Peroral endoscopic myotomy

INTERVENTIONS:
Procedure: Peroral endoscopic myotomy — Patients will be hospitalized for 24 hours before procedure or at the day of procedure (depending on preference of each center). Procedures will be performed always using carbon dioxide insufflation and whenever possible under general anesthesia with endotracheal intubation by anesthesiologist recommendations. The procedure will begin after general endoscopic evaluation of the Zenker's diverticulum and esophagus. An incision of the bridge between the Zenker's diverticulum and the esophagus will be done using procedure as peroral endoscopic myotomy. All the procedures will be documented with photographs or videorecordings.
  Other Names: Z-POEM
  Arms: Investigational procedure
Procedure: Flexible endoscopic septotomy — Patients will be hospitalized for 24 hours before procedure or at the day of procedure (depending on preference of each center). Procedures will be performed always using carbon dioxide insufflation and whenever possible under general anesthesia with endotracheal intubation by anesthesiologist recommendations. The procedure will begin after general endoscopic evaluation of the Zenker's diverticulum and esophagus. An incision of the bridge between the Zenker's diverticulum and the esophagus will be done using procedure as flexible endoscopy septotomy. All the procedures will be documented with photographs or videorecordings.
  Arms: Standard procedure

SUMMARY:
The Zenker's or pharyngo-esophageal diverticulum is an acquired sac-like outpouching of the mucosa and submucosa layers located dorsally at the pharyngoesophageal junction through Killian's dehiscence. It is the most common type of oesophageal diverticula and typically occurs in middle-aged and elderly patients. Patients have a significantly reduced quality of life index and numerous complications.

Treatment is recommended for symptomatic patients and considering the aetiopathogenesis of the disease demands myotomy of the cricopharyngeal muscle. Myotomy may be pursued through either open surgical or endoscopic techniques.

There is a novel technique, called the peroral endoscopic myotomy (Z-POEM) for treatment of Zenker's diverticulum.

The ZIPPY trial designed as prospective, international, multicenter, double-blind, randomized study which will be carried out by experienced endoscopists. The aim of this study will be to evaluate the results of Zenker's diverticulum treatment using peroral endoscopic myotomy and to compare its efficacy and safety to flexible endoscopy septotomy. Patients at least 18 years old with symptomatic Zenker's diverticulum diagnosed on the basis of endoscopic and radiological examinations will be enrolled.

DETAILED DESCRIPTION:
Participants will be randomized into one of two groups: (I) Z-POEM, (II) flexible endoscopic septotomy. Patients with clinical failure will be offered other method of treatment and will be included to observational cohort. The study has been approved by a local bioethics committee

ELIGIBILITY:
Inclusion Criteria:

1. Males and females who are 18 years of age and older and are able to comprehend instructions and follow the study procedures and are willing to sign an Informed Consent Form (ICF).
2. Patients with symptomatic Zenker's Diverticulum.
3. Confirmed diagnosis of Zenker's Diverticulum based on endoscopic and radiological examinations.
4. Size of Zenker's Diverticulum in the range of 1,5 to 4 cm on radiological examinations.

Exclusion Criteria:

1. Lack of written consent for participation in the study.
2. Size of Zenker's Diverticulum <1,5 cm or >4 cm on radiological examination.
3. Active cancer.
4. Esophageal stricture.
5. Eosinophilic esophagitis (EoE).
6. Pre-cancerous changes in the esophagus.
7. Previous surgical or endoscopic treatment of Zenker's Diverticulum.
8. Presence of chewing deficiencies and/or neurogenic dysphagia.
9. Presence of other esophageal motility disorders e.g. achalasia and/or spastic motility disorders.
10. Severe systemic diseases which are contraindication to general sedation.
11. Severe coagulopathy.
12. Pregnancy and breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Rate of procedural technical success defined as completion of all steps of Z-POEM including complete cricopharyngeus myotomy. | 3 Months
Rate of short-term clinical success defined as complete or near complete resolution of postprocedure dysphagia and other related symptoms (regurgitation, halitosis, cough, hoarseness, weight loss, episodes of aspiration pneumonia). | 3 Months

SECONDARY OUTCOMES:
Rate of long-term clinical success defined as lack of recurrence during 24 months follow-up | 24 Months
Assessment of clinical symptoms severity measured with the scale EAT-10 | 24 Months
Assessment of clinical symptoms severity measured with the scale FOSS | 24 Months
Percentage of adverse events with graded severity. | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Michal Filip Kaminski, MD, PhD, Principal Investigator — Professor of Department of Cancer Prevention and Center of Oncology Institute
Locations (1):
- The Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PubMed Identifier — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6441918/
- See also: PubMed Identifier — https://pubmed.ncbi.nlm.nih.gov/31082393/
- See also: PubMed Identifier — https://pubmed.ncbi.nlm.nih.gov/30453378/
- See also: MedlinePlus — https://medlineplus.gov/endoscopy.html